CLINICAL TRIAL: NCT04032275
Title: Correlation Between Virus and Biochemical Characteristics and Liver Histological Damage in Untreated Patients With Chronic HBV Infection
Brief Title: Correlation Between Virus and Biochemical Characteristics and Liver Histological Damage in Untreated Chronic HBV Infection
Status: Completed | Type: Observational
Sponsor: Beijing Ditan Hospital (Other)
Responsible Party: Principal Investigator, Yao Xie, Head of liver diseases center, Beijing Ditan Hospital
Other Study IDs: DTXY020
Record Dates: First submitted 2019-07-20; First posted 2019-07-25 (Actual); Last update posted 2019-07-25 (Actual); Status verified 2019-07

CONDITIONS: Chronic Hepatitis B
Keywords: chronic hepatitis B; HBV; HBsAg; HBeAg; HBV DNA; histological examination
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Untreated chronic HBV infected person group: Enrolled in the Department of Hepatology, Beijing Ditan Hospital, Capital Medical University, Department of Liver Histology, Department of Hepatology, Chronic HBV HBV infection.
  Interventions: Other: Chronic hepatitis B infection

INTERVENTIONS:
Other: Chronic hepatitis B infection — Chronic hepatitis B infection patients

SUMMARY:
This study is a retrospective study. Enrollment study. Enrolled in the Department of Hepatology, Beijing Ditan Hospital, Capital Medical University, Department of Liver Histology, Department of Hepatology, Chronic HBV HBV infection. The data collected included patient gender, . The data collected included patient gender, . The data collected included the patient's gender, age, HBV age of infection, past family history, etc., the age of the collected subjects, the current family history, etc., the liver histopathological diagnosis information collected in the group, and the liver disease examination Clinical toxicities and indicators, including serological diagnostic information, clinical toxicities and indicators for liver disease tests, including serological diagnostic information, clinical toxicities and indicators for liver disease tests, including serum HBV DNA HBV DNAHBV DNAHBV DNA HBV DNA content, HBsAg/HBsAg/HBsAg/HBsAg/anti-HBsHBsHBs, HBeAg/HBeAg/HBeAg/HBeAg/HBeAg/anti-HBe content, biochemical indicators coagulation function and routine data. Content, biochemical indicators, coagulation function and routine data. Content, biochemical indicators, coagulation function and routine data. Observe patient demographic data, HBV DNA HBV DNAHBV DNAHBV DNA HBV DNA content, HBsAg/HBsAg/HBsAg/HBsAg/HBsAg/anti-HBsHBsHBs, HBeAg/HBeAg/HBeAg/HBeAg/HBeAg/HBeAg/anti-HBe HBe content, biochemical indicators, coagulation Correlation between function and routine, coagulation function and conventional indicators and liver histological changes. Explore the relevance of effective diagnosis of liver changes. To explore the characteristics of clinical indicators that can effectively diagnose liver histopathological changes, and to provide clinical indicators for patients with chronic hepatitis B to receive timely treatment of histopathological changes, and provide important evidence for patients with chronic hepatitis B to receive timely treatment.

DETAILED DESCRIPTION:
This study is a retrospective study. Enrollment study. Enrolled in the Department of Hepatology, Beijing Ditan Hospital, Capital Medical University, Department of Liver Histology, Department of Hepatology, Chronic HBV HBV infection. The data collected included patient gender, . The data collected included patient gender, . The data collected included the patient's gender, age, HBV age of infection, past family history, etc., the age of the collected subjects, the current family history, etc., the liver histopathological diagnosis information collected in the group, and the liver disease examination Clinical toxicities and indicators, including serological diagnostic information, clinical toxicities and indicators for liver disease tests, including serological diagnostic information, clinical toxicities and indicators for liver disease tests, including serum HBV DNA HBV DNAHBV DNAHBV DNA HBV DNA content, HBsAg/HBsAg/HBsAg/HBsAg/anti-HBsHBsHBs, HBeAg/HBeAg/HBeAg/HBeAg/HBeAg/anti-HBe content, biochemical indicators coagulation function and routine data. Content, biochemical indicators, coagulation function and routine data. Content, biochemical indicators, coagulation function and routine data. Observe patient demographic data, HBV DNA HBV DNAHBV DNAHBV DNA HBV DNA content, HBsAg/HBsAg/HBsAg/HBsAg/HBsAg/anti-HBsHBsHBs, HBeAg/HBeAg/HBeAg/HBeAg/HBeAg/HBeAg/anti-HBe HBe content, biochemical indicators, coagulation Correlation between function and routine, coagulation function and conventional indicators and liver histological changes. Explore the relevance of effective diagnosis of liver changes. To explore the characteristics of clinical indicators that can effectively diagnose liver histopathological changes, and to provide clinical indicators for patients with chronic hepatitis B to receive timely treatment of histopathological changes, and provide important evidence for patients with chronic hepatitis B to receive timely treatment.

ELIGIBILITY:
Inclusion Criteria:

* 1) Age between 18 and over 65;
* 2) gender is not limited;
* 3) Patients with chronic HBVHBVHBV infection: all meet the diagnostic criteria of China's Guidelines for the Prevention and Treatment of Chronic Hepatitis B (: all meet the diagnostic criteria for the Chinese Guidelines for the Prevention and Treatment of Chronic Hepatitis B (2015), HBsAg HBsAg HBsAg positive for 6 months Month;
* 4) Sign the written informed consent.Exclusion Criteria:

Exclusion Criteria:

* 1) Combine other hepatitis viruses (HCV (HCV, HDV, HDV) infection;
* 2) autoimmune liver disease;
* 3) HIVHIV HIV infection;
* 4) long-term alcohol abuse and / or other liver damage drugs;
* 5) mental illness;
* 6) Evidence of liver tumors (cancer or AFP AFP>100 ng/ml 100 ng/ml 100 ng/ml 100 ng/ml);
* 7) decompensated cirrhosis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic HBVHBVHBV infection: all meet the diagnostic criteria of China's Guidelines for the Prevention and Treatment of Chronic Hepatitis B (: all meet the diagnostic criteria for the Chinese Guidelines for the Prevention and Treatment of Chronic Hepatitis B (2015), HBsAg HBsAg HBsAg positive for 6 months Month;
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
the diagnostic ability of clinical indicators | 6 months
  Clinical indicators characterize the diagnostic ability of liver histology inflammation and fibrosis

CONTACTS AND LOCATIONS:
Overall Officials: Yao Xie, Doctor, Principal Investigator — Beijing Ditan Hospital, Beijing, China
Locations (1):
- liver disease center, Beijing Ditan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No